CLINICAL TRIAL: NCT00425750
Title: Phase II Trial of Combination Weekly Bortezomib (VELCADE) and Docetaxel (TAXOTERE) in Patients With Recurrent and/ or Metastatic Head and Neck Squamous Cell Carcinoma (HNSCC)
Brief Title: Bortezomib and Docetaxel in Treating Patients With Recurrent or Metastatic Head and Neck Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Vanderbilt-Ingram Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Principal Investigator, Barbara Murphy, Professor of Medicine; Director, Cancer Supportive Care Program; Director, Head and Neck Research Program; Medical Oncologist, Vanderbilt-Ingram Cancer Center
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: VICC HN 0501; P30CA068485 (NIH); VU-VICC-HN-0501; MILLENIUM-X05170; VU-VICC-IRB-050183
Record Dates: First submitted 2007-01-19; First posted 2007-01-23 (Estimated); Results first posted 2011-04-04 (Estimated); Last update posted 2011-11-16 (Estimated); Status verified 2011-11

CONDITIONS: Head and Neck Cancer
Keywords: stage IV squamous cell carcinoma of the lip and oral cavity; recurrent squamous cell carcinoma of the lip and oral cavity; stage IV squamous cell carcinoma of the oropharynx; recurrent squamous cell carcinoma of the oropharynx; stage IV squamous cell carcinoma of the hypopharynx; recurrent squamous cell carcinoma of the hypopharynx; stage IV squamous cell carcinoma of the larynx; recurrent squamous cell carcinoma of the larynx
MeSH Terms: conditions — Head and Neck Neoplasms; Squamous Cell Carcinoma of Head and Neck | interventions — Bortezomib; Docetaxel

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Treatment (Experimental): Docetaxel (40 mg/m2) IV Infusion over 30 minutes every 3 weeks (Day 1 and 8 of 21 day cycle)except the first dose is held on Day 1 of Cycle 1.
  Bortezomib (1.6mg/m2) IV 3-5 second push every 3 weeks (Day 1 and 8 of 21 day cycle).Bortezomib is given as a single agent only on Day 1 of Cycle 1.
  Interventions: Drug: bortezomib; Drug: docetaxel; Other: laboratory biomarker analysis; Other: pharmacological study

INTERVENTIONS:
Drug: bortezomib — 1.6 mg/m2 through a vein on days 1 and 8 of a 21-day cycle. The first dose is given as a single agent only on Day 1 of Cycle 1.
Drug: docetaxel — 40 mg/m2 through a vein on days 1 and 8 of a 21-day cycle except the first dose is held only on Day 1 of Cycle 1.
Other: laboratory biomarker analysis — Tissue and blood collection.
Other: pharmacological study — Blood collection.

SUMMARY:
RATIONALE: Bortezomib may stop the growth of tumor cells by blocking some of the enzymes needed for cell growth. It may also stop the growth of tumor cells by blocking blood flow to the tumor. Drugs used in chemotherapy, such as docetaxel, work in different ways to stop the growth of tumor cells, either by killing the cells or by stopping them from dividing. Giving bortezomib together with docetaxel may kill more tumor cells.

PURPOSE: This phase II trial is studying how well giving bortezomib together with docetaxel works in treating patients with recurrent or metastatic head and neck cancer.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* Determine the overall response rate in patients with recurrent and/or metastatic squamous cell carcinoma of the head and neck treated with bortezomib and docetaxel.

Secondary

* Determine the time to progression in patients treated with this regimen.
* Determine the toxicity of this regimen.
* Determine the duration of response in patients treated with this regimen.
* Determine the overall survival and progression-free survival of these patients.
* Determine 20S proteasome inhibition in peripheral blood mononuclear cells (PBMC) from these patients.
* Determine the effect of bortezomib on NF-kB pathway in PBMC and serum samples.
* Identify biomarkers of clinical response to bortezomib and docetaxel in PBMC and serum.
* Determine quality of life, symptom burden, and physical function outcome in patients treated with this regimen.

OUTLINE: This is a prospective, open-label, nonrandomized study.

Patients receive docetaxel* IV over 30 minutes and bortezomib IV on days 1 and 8. Courses repeat every 28 days in the absence of disease progression or unacceptable toxicity.

NOTE: *Docetaxel is not administered on day 1 of course 1.

Blood samples are collected at baseline, after bortezomib administration on day 1 of course 1, and at the completion of treatment. The pharmacodynamics and pharmacogenomics of bortezomib are assessed in peripheral blood mononuclear cells (PBMC) and serum.

After completion of study treatment, patients are followed every 6 weeks for 1 year and then every 3 months thereafter.

PROJECTED ACCRUAL: A total of 50 patients will be accrued for this study.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Diagnosis of squamous cell carcinoma of the oral cavity, oropharynx, hypopharynx, or larynx

  * Recurrent or metastatic disease
* Measurable disease
* Not a candidate for curative therapy

PATIENT CHARACTERISTICS:

* ECOG performance status 0-2
* Absolute neutrophil count ≥ 1,500/mm³
* Hemoglobin ≥ 8.0 g/dL
* Platelet count ≥ 100,000/mm³
* AST, ALT, and alkaline phosphatase (AP) meeting 1 of the following criteria:

  * AP normal AND AST and ALT ≤ 5 times upper limit of normal (ULN)
  * AP ≤ 2.5 times ULN AND AST and ALT ≤ 1.5 times ULN
  * AP ≤ 5 times ULN AND AST and ALT normal
* Bilirubin normal
* Creatinine clearance ≤ 2.0 mg/dL
* No peripheral neuropathy ≥ grade 2 within the past 28 days
* No myocardial infarction within the past 6 months
* No New York Heart Association class III or IV heart failure
* No uncontrolled angina
* No severe uncontrolled ventricular arrhythmias
* No electrocardiographic evidence of acute ischemia or active conduction system abnormalities
* No known hypersensitivity to bortezomib, boron, or mannitol
* No known severe hypersensitivity reaction to docetaxel or other drugs formulated with polysorbate 80
* No serious medical or psychiatric illness that would preclude study participation
* No other malignancy within the past 3 years except for early-stage nonmelanomatous skin cancer, carcinoma in situ of the cervix, or early-stage prostate cancer
* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective contraception during and for ≥ 3 months after completion of study treatment

PRIOR CONCURRENT THERAPY:

* No prior chemotherapy for recurrent or metastatic disease
* At least 28 days since prior and no other concurrent investigational drugs
* No other concurrent anticancer therapy
* No other concurrent chemotherapy
* No concurrent complementary or herbal medicine
* No concurrent filgrastim (G-CSF) or sargramostim (GM-CSF)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Actual)
Dates: Start 2005-08; Primary Completion 2009-06 (Actual); Study Completion 2009-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Barbara Murphy, MD, Study Chair — Vanderbilt-Ingram Cancer Center
Locations (7):
- United States (7):
  - Jennie Stuart Medical Center, Hopkinsville, Kentucky
  - Purchase Cancer Group - Paducah, Paducah, Kentucky
  - Tennessee Plateau Oncology - Crossville, Crossville, Tennessee
  - West Tennessee Cancer Center at Jackson-Madison County General Hospital, Jackson, Tennessee
  - Baptist Regional Cancer Center at Baptist Riverside, Knoxville, Tennessee
  - MBCCOP - Meharry Medical College - Nashville, Nashville, Tennessee
  - Vanderbilt-Ingram Cancer Center, Nashville, Tennessee

REFERENCES:
- [Result] Chung CH, Aulino J, Muldowney NJ, Hatakeyama H, Baumann J, Burkey B, Netterville J, Sinard R, Yarbrough WG, Cmelak AJ, Slebos RJ, Shyr Y, Parker J, Gilbert J, Murphy BA. Nuclear factor-kappa B pathway and response in a phase II trial of bortezomib and docetaxel in patients with recurrent and/or metastatic head and neck squamous cell carcinoma. Ann Oncol. 2010 Apr;21(4):864-870. doi: 10.1093/annonc/mdp390. Epub 2009 Oct 22. PMID 19850643
- [Derived] Chung CH, Lee JW, Slebos RJ, Howard JD, Perez J, Kang H, Fertig EJ, Considine M, Gilbert J, Murphy BA, Nallur S, Paranjape T, Jordan RC, Garcia J, Burtness B, Forastiere AA, Weidhaas JB. A 3'-UTR KRAS-variant is associated with cisplatin resistance in patients with recurrent and/or metastatic head and neck squamous cell carcinoma. Ann Oncol. 2014 Nov;25(11):2230-2236. doi: 10.1093/annonc/mdu367. Epub 2014 Jul 31. PMID 25081901

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This study was open to accrual from 8/25/2005 through 5/20/2008.
Pre-assignment Details: Twenty-seven patients consented, two of which were ineligible.
Groups:
- Bortezomib; Docetaxel: Docetaxel will be given first at 40 mg/m2 IV on days 1 and 8 of a 21-day cycle except the first dose is held only on Day 1 of Cycle 1. Immediately afterwards, Bortezomib will be given at 1.6 mg/m2 IV on days 1 and 8 of a 21-day cycle. The first dose is given as a single agent only on Day 1 of Cycle 1.
Period: Overall Study
Arm/Group | Bortezomib; Docetaxel
Started | 25
Completed | 0
Not Completed | 25
Not completed — Death | 1
Not completed — Withdrawal by Subject | 3
Not completed — Adverse Event | 3
Not completed — Progression of disease | 18

BASELINE CHARACTERISTICS:
Arm/Group | Bortezomib; Docetaxel
Number analyzed (Participants) | 25
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 21
  >=65 years | 4
Age Continuous [Mean (Standard Deviation); unit: years] | 55 (1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 7
  Male | 18
Region of Enrollment [Number; unit: participants]
  United States | 25

OUTCOME MEASURES:

1. Primary Outcome: Patient Response to Treatment
Description: Progressive disease (PD): >=20% increase in sum of longest diameter (LD) of target lesion(s), taking as reference smallest sum LD recorded since treatment started. Complete response (CR): disappearance of all target lesions. Partial response (PR): >=30% decrease in sum of LD of target lesion(s), taking as reference baseline sum LD. Stable disease (SD): neither sufficient shrinkage to qualify as PR nor sufficient increase to qualify as PD.
Time Frame: 7.55 months (average duration, on study to off study)
Measure: Number; unit: participants
Arm/Group | Bortezomib; Docetaxel
Number analyzed (Participants) | 25
participants
  Partial Response | 1
  Progressive Disease | 10
  Stable Disease | 10
  Not Evaluable | 4

2. Secondary Outcome: Overall Survival
Description: Median survival time of patients, calculated as on-study date to date of death or off-study date (censored)
Time Frame: 7.55 months (average duration, on study to off study)
Measure: Median (95% Confidence Interval); unit: Month
Arm/Group | Bortezomib; Docetaxel
Number analyzed (Participants) | 25
Month | 5.13 [3.71 to 9.76]

3. Secondary Outcome: Progression-free Survival
Description: Median duration of survival without disease progression, calculated as on-study date to date of progression or date of death (censored) or off-study date (censored)
Time Frame: 7.55 months (average duration, on study to off study)
Measure: Median (95% Confidence Interval); unit: Month
Arm/Group | Bortezomib; Docetaxel
Number analyzed (Participants) | 25
Month | 2.27 [1.61 to 4.70]

ADVERSE EVENTS:
Arm/Group | Bortezomib; Docetaxel
Serious Adverse Events (participants affected / at risk) | 11/25
Other Adverse Events (participants affected / at risk) | 0/25
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Bortezomib; Docetaxel (N=25)
Death (General disorders) | 2 (2)
Vomitting (Gastrointestinal disorders) | 2 (2)
Hypercalcemia (Metabolism and nutrition disorders) | 1 (1)
Seizure (Nervous system disorders) | 1 (1)
Diarrhea (Gastrointestinal disorders) | 1 (1)
Dry mouth (Gastrointestinal disorders) | 1 (1)
Mucositis (Gastrointestinal disorders) | 1 (1)
Nausea (Gastrointestinal disorders) | 1 (1)
Hemorrhage, GI (Gastrointestinal disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes